CLINICAL TRIAL: NCT06662942
Title: A Double Blind Placebo-controlled Trial of StrataMGT for the Management of Vulvar Lichen Sclerosus Symptoms.
Brief Title: StrataMGT in the Reduction of Vulvar Lichen Sclerosus (LS) Symptoms
Acronym: LS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew T. Goldstein, MD (Other)
Collaborators: Stratpharma AG (Industry)
Responsible Party: Sponsor-Investigator, Andrew T. Goldstein, MD, Principal Investigator, Center for Vulvovaginal Disorders
Organization: Center for Vulvovaginal Disorders (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVVD005; 24-02-237 (Other: BRANY IRB)
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: StrataMGT
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (Active Comparator): StrataMGT® is a semi-permeable, non-resorbable and self-drying gel. StrataMGT® contains no steroids, hormones, alcohol, parabens or fragrances. StrataMGT® gel is bacteriostatic, inert, and is manufactured in compliance with good manufacturing practices (GMPs), 21CFR210 and 211.
  Interventions: Drug: StrataMGT
- Placebo (Placebo Comparator): This arm will be a sterile, transparent, water-soluble lubricating jelly that is not silicone-based.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: StrataMGT — StrataMGT® is a semi-permeable, non-resorbable and self-drying gel. StrataMGT® contains no steroids, hormones, alcohol, parabens or fragrances. StrataMGT® gel is bacteriostatic, inert, and is manufactured in compliance with good manufacturing practices (GMPs), 21CFR210 and 211.
  Arms: Investigational product
Drug: Placebo — The placebo is a sterile, transparent, water-soluble lubricating jelly that is not silicone-based. It will be applied topically to the vulvar skin.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of StrataMGT for the management of vulvar lichen sclerosus symptoms.

DETAILED DESCRIPTION:
This will be a randomized double-blind placebo-controlled trial to evaluate the efficacy and safety of StrataMGT for the management of the symptoms of vulvar lichen sclerosus. Up to 100 patients with a diagnosis of biopsy proven vulvar lichen sclerosus will be recruited from two centers. This study will consist of a two-week screening period and a 12-week treatment period. At the beginning of the screening period, a vulvoscopy will be performed at the screening visit and after the 12-week treatment period to rule out vulvar intrepithelial neoplasia (VIN) or carcinoma. All eligible patients will be randomized to receive either placebo gel or treatments with the investigation product, StrataMGT TM 1:1 ratio.

The primary efficacy endpoint will be change in score on the Vulvar Quality of Life Index 11 (VQLI).

Secondary efficacy endpoints will be the Skindex 29, and the Clinical Lichen Sclerosus Scoring Scale (CLISSCO).

All adverse events will be recorded, including serious adverse events. A physical examination will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years or older.
* With a diagnosis of biopsy proven vulvar lichen sclerosus.
* Signed written informed consent.
* Willingness and ability to comply with the study requirements.
* Subject must have a score of 10 or greater in the VQLI at screening.
* Must be on a stable regimen of topical corticosteroids or topical calcineurin inhibitor for at least 2 months prior to the screening visit.
* Women currently on a stable regimen of intravaginal estrogen therapy for at least 2 months may remain on the estrogen therapy throughout the study.
* Women currently using topical estrogen therapy on the vulva must stop two weeks prior to enrolling in the study.
* Women must have a culture negative for candidiasis or bacterial vaginosis at screening.

Exclusion Criteria:

* Who are immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease.
* Who suffer from a topical or systemic infections (bacterial, viral or fungal) at the time of screening. Subjects who screen positive for either candidiasis or bacterial vaginosis at the screening visit may be treated and retested and may participate if the confirmatory test after treatment is negative. Any vulvovaginal infections during their participation in the study will be considered an adverse event. The subject will then stop the study IP and will be treated for the infection and may resume use of the IP 3 days after the last dose of medication for the infection. They will be discontinued from the study if they have two infections during the study.
* Who have been diagnosed with lichen planus, psoriasis, intraepithelial neoplasia, or carcinoma of the vulva.
* Who had received an investigational drug within four weeks prior to the study or who intend to use other investigational drugs during the course of this study.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Who have a history of substance abuse or any factor, which limits the subject's ability to cooperate with the study procedures.
* Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions or are not willing to attend regularly scheduled visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Vulvar Quality of Life Index 11 (VQLI) | throughout the study, averaging 3.5 months
  The VQLI is used to "assess symptomatic, psychosexual and physical aspects of vulvar disease" [1] using the following scale: Very Much, A Lot, A Little, and Not At All. The questionnaire consists of 15 questions.

SECONDARY OUTCOMES:
Skindex 29 | throughout the study, averaging 3.5 months
  The Skindex 29 is a subjective survey used to assess which skin conditions have bothered a patient the most on the following scale: All the time, often, sometimes, rarely, and never. The survey consists of 30 questions.
Clinical Scoring System for Vulvar Lichen Sclerosus | throughout the study, averaging 3.5 months
  The Clinical Scoring System for Vulvar Lichen Sclerosus is a subjective and objective survey filled out by the patient and provider. It is used to assess the patient's severity of subjective symptoms and the provider's interpretation of the severity of visible symptoms associated with vulvar LS.

CONTACTS AND LOCATIONS:
Overall Officials: Chailee Moss, MD, Study Director — Centers for Vulvovaginal Disorders, DC; Jill Krapf, MD, Study Director — Centers for Vulvovaginal Disorders, FL
Locations (3):
- United States (3):
  - Centers for Vulvovaginal Disorders, DC, Washington D.C., District of Columbia
  - Centers for Vulvovaginal Disorders, FL, Tampa, Florida
  - Centers for Vulvovaginal Disorders, NY, New York, New York

IPD SHARING:
Plan to Share IPD: No